CLINICAL TRIAL: NCT00000446
Title: Sertraline Treatment in Comorbid Post-Traumatic Stress Disorder and Alcoholism
Brief Title: Drug Treatment for Alcoholics With Post-Traumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAABRA10761
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-04

CONDITIONS: Alcoholism; Post-Traumatic Stress Disorder
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Sertraline

INTERVENTIONS:
Drug: sertraline (Zoloft)

SUMMARY:
This study will investigate the use of sertraline (Zoloft) to decrease alcohol consumption and crime-related post-traumatic stress disorder in those individuals with both disorders. This will be a 12-week, placebo-controlled, double-blind outpatient trial.

All subjects will receive cognitive behavioral therapy in addition to a placebo or sertraline. Comprehensive evaluation will be done at study entry; treatment termination; and 6, 9, and 12 months after study entry.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for alcohol abuse or dependence and post-traumatic stress disorder.
* Laboratory tests for blood and urinalysis must be within normal limits.
* Must be clearly motivated to obtain benefit from treatment and keep appointments for study visits and therapy sessions.
* Females who use an acceptable method of birth control, are sterilized, or are at least 2 years post-menopausal.

Exclusion Criteria:

* Have a diagnosis of schizophrenia, bipolar affective disorder, dissociative identity disorder, eating disorder, substance dependence in the last 60 days.
* Currently suicidal.
* Medical reasons not to receive drug therapy.
* Allergy or hypersensitivity to selective serotonin inhibitor antidepressants.
* Significant hematological, endocrine, cardiovascular, renal, hepatic, neurological, or gastrointestinal disease.
* Liver function test greater than 2 times the normal level
* Require ongoing therapy with another psychoactive drug during the study period.
* Females who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2000-12

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Behavioral Science, Medical University of South Carolina, Charleston, South Carolina, United States